CLINICAL TRIAL: NCT01623856
Title: Observational - Candidate Gene Variants and Childhood/Adolescent Non-Hodgkin Lymphoma: A Preliminary Investigation
Brief Title: Studying Genes Associated With Non-Hodgkin Lymphoma in Young Patients
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANHL12B1; NCI-2012-01975 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-06-15; First posted 2012-06-20 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Childhood Burkitt Lymphoma; Childhood Lymphoblastic Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: DNA samples are analyzed by single nucleotide polymorphism and genotyped by fluorogenic polymerase chain reaction (PCR)-based allelic discrimination (Taqman) assays using the ABI Prism 7900HT reverse transcriptase (RT)-PCR system.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research studies genes associated with non-Hodgkin lymphoma in young patients. Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. To conduct a preliminary investigation of the effects of loci strongly and consistently associated in prior genome-wide association studies (GWAS) and validation studies of childhood/adolescent acute lymphoblastic leukemia (ALL), adult non-Hodgkin lymphoma (NHL), autoimmune diseases, and atopic diseases on the risk of NHL (lymphoblastic and Burkitt lymphomas) in children and adolescents.

OUTLINE:

DNA samples are analyzed by single nucleotide polymorphism and genotyped by fluorogenic polymerase chain reaction (PCR)-based allelic discrimination (Taqman) assays using the ABI Prism 7900HT reverse transcriptase (RT)-PCR system.

ELIGIBILITY:
Inclusion Criteria:

* Slides and/or other available specimens from patients diagnosed with lymphoblastic lymphoma (LL) or Burkitt lymphoma ( BL) enrolled on the Children Oncology Group (COG) protocols 5961, A5971, and ANHL01P1 collected at the time of diagnosis and currently housed at the Biopathology Center at Nationwide Children's Hospital

  * Samples from non-Hispanic white patients
* DNA samples from 384 healthy, anonymous, non-Hispanic white blood donors used as controls
* See Disease Characteristics
* Not specified

Max Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients diagnosed with lymphoblastic lymphoma (LL) or Burkitt lymphoma ( BL) enrolled on the Children Oncology Group (COG) protocols 5961, A5971, or ANHL01P1.
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2012-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Potential deviations from Hardy-Weinberg Equilibrium (HWE) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Amy Linabery, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States